CLINICAL TRIAL: NCT04626856
Title: Evaluation of the Safety and Preliminary Immunogenicity of Inactivated Rotavirus Vaccine (Vero Cell) in Healthy Population: a Randomized, Double-blind, Placebo Parallel-controlled Phase I Clinical Trial
Brief Title: Safety and Preliminary Immunogenicity Study of Inactivated Vaccine for Prevention of Rotavirus Infection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Henan Provincal Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Li Hongjun, PI, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AF/SC-08/03.0
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Rotavirus Infection
MeSH Terms: conditions — Rotavirus Infections | interventions — Appointments and Schedules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Low dosage in adults (Experimental): Low dosage Inactivated Rotavirus vaccine (Vero cell) in adults aged 18-49 years old on day 0, 28
  Interventions: Biological: Low dosage IRV on a 0- and 28-day schedule
- Medium dosage in adults (Experimental): Medium dosage Inactivated Rotavirus vaccine (Vero cell) in adults aged 18-49 years old on day 0, 28
  Interventions: Biological: Medium dosage IRV on a 0- and 28-day schedule
- High dosage in adults (Experimental): High dosage Inactivated Rotavirus vaccine (Vero cell) in adults aged 18-49 years old on day 0, 28
  Interventions: Biological: High dosage IRV on a 0- and 28-day schedule
- Low dosage in adolescents (Experimental): Low dosage Inactivated Rotavirus vaccine (Vero cell) in adolescents aged 6-17 years old on day 0, 28
  Interventions: Biological: Low dosage IRV on a 0- and 28-day schedule
- Medium dosage in adolescents (Experimental): Medium dosage Inactivated Rotavirus vaccine (Vero cell) in adolescents aged 6-17 years old on day 0, 28
  Interventions: Biological: Medium dosage IRV on a 0- and 28-day schedule
- High dosage in adolescents (Experimental): High dosage Inactivated Rotavirus vaccine (Vero cell) in adolescents aged 6-17 years old on day 0, 28
  Interventions: Biological: High dosage IRV on a 0- and 28-day schedule
- Low dosage in infants (7-71 months old) (Experimental): Low dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 7-71 months old on day 0, 28
  Interventions: Biological: Low dosage IRV on a 0- and 28-day schedule
- Medium dosage in infants (7-71 months old) (Experimental): Medium dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 7-71 months old on day 0, 28
  Interventions: Biological: Medium dosage IRV on a 0- and 28-day schedule
- High dosage in infants (7-71 months old) (Experimental): High dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 7-71 months old on day 0, 28
  Interventions: Biological: High dosage IRV on a 0- and 28-day schedule
- Low dosage in infants (2-6 months old, two-dose) (Experimental): Low dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 2-6 months old on day 0, 28
  Interventions: Biological: Low dosage IRV on a 0- and 28-day schedule
- Medium dosage in infants (2-6 months old, two-dose) (Experimental): Medium dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 2-6 months old on day 0, 28
  Interventions: Biological: Medium dosage IRV on a 0- and 28-day schedule
- High dosage in infants (2-6 months old, two-dose) (Experimental): High dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 2-6 months old on day 0, 28
  Interventions: Biological: High dosage IRV on a 0- and 28-day schedule
- Low dosage in infants (2-6 months old, three-dose) (Experimental): Low dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 2-6 months old on day 0, 28, 56
  Interventions: Biological: Low dosage IRV on a 0- , 28- and 56-day schedule
- Medium dosage in infants (2-6 months old, three-dose) (Experimental): Medium dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 2-6 months old on day 0, 28, 56
  Interventions: Biological: Medium dosage IRV on a 0- , 28- and 56-day schedule
- High dosage in infants (2-6 months old, three-dose) (Experimental): High dosage Inactivated Rotavirus vaccine (Vero cell) in infants aged 2-6 months old on day 0, 28, 56
  Interventions: Biological: High dosage IRV on a 0- , 28- and 56-day schedule
- Placebo on day 0, 28 (Placebo Comparator): Two doses of placebo at the vaccination schedule of day 0,28
  Interventions: Biological: Placebo on day 0, 28
- Placebo on day 0, 28, 56 (Placebo Comparator): Three doses of placebo at the vaccination schedule of day 0, 28,56
  Interventions: Biological: Placebo on day 0, 28, 56

INTERVENTIONS:
Biological: Low dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 80EU/0.5ml on day 0, 28
  Arms: Low dosage in adults
Biological: Medium dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 160EU/0.5ml on day 0, 28
  Arms: Medium dosage in adults
Biological: High dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 320EU/0.5ml on day 0,28
  Arms: High dosage in adults
Biological: Low dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 80EU/0.5ml on day 0,28
  Arms: Low dosage in adolescents
Biological: Medium dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 160EU/0.5ml on day 0,28
  Arms: Medium dosage in adolescents
Biological: High dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 320EU/0.5ml on day 0,28
  Arms: High dosage in adolescents
Biological: Low dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 80EU/0.5ml on day 0,28
  Arms: Low dosage in infants (7-71 months old)
Biological: Medium dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 160EU/0.5ml on day 0,28
  Arms: Medium dosage in infants (7-71 months old)
Biological: High dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 320EU/0.5ml on day 0,28
  Arms: High dosage in infants (7-71 months old)
Biological: Low dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 80EU/0.5ml on day 0,28
  Arms: Low dosage in infants (2-6 months old, two-dose)
Biological: Medium dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 160EU/0.5ml on day 0,28
  Arms: Medium dosage in infants (2-6 months old, two-dose)
Biological: High dosage IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 320EU/0.5ml on day 0,28
  Arms: High dosage in infants (2-6 months old, two-dose)
Biological: Low dosage IRV on a 0- , 28- and 56-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 80EU/0.5ml on day 0,28,56
  Arms: Low dosage in infants (2-6 months old, three-dose)
Biological: Medium dosage IRV on a 0- , 28- and 56-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 160EU/0.5ml on day 0,28,56
  Arms: Medium dosage in infants (2-6 months old, three-dose)
Biological: High dosage IRV on a 0- , 28- and 56-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 320EU/0.5ml on day 0,28,56
  Arms: High dosage in infants (2-6 months old, three-dose)
Biological: Placebo on day 0, 28 — Two doses of placebo at the vaccination schedule of day 0,28
  Arms: Placebo on day 0, 28
Biological: Placebo on day 0, 28, 56 — Three doses of placebo at the vaccination schedule of day 0, 28,56
  Arms: Placebo on day 0, 28, 56

SUMMARY:
This study is a randomized, double-blinded, placebo-controlled, Phase 1, dose-escalation study to evaluate the safety, reactogenicity and immunogenicity of Inactivated Rotavirus Vaccine (IRV) performed in healthy adult (aged 18-49 years), adolescent (aged 6-17 years) and infant subjects (aged 2-71 months). Primary objectives of the clinical trial include assessing the safety and tolerability of IRV given at two and three dose levels and comparing the safety and tolerability of IRV after each vaccination, between dosage groups, and by pre-vaccination rotavirus immune status. Secondary objective of the clinical trial is immunogenicity evaluation after each vaccination, between dosage groups, and by pre-vaccination rotavirus immune status.

DETAILED DESCRIPTION:
This clinical trial aimed to evaluate safety and immunogenicity effect of IRV（Vero cell）in Chinese healthy adults, adolescents and infants. The subjects were divided into 5 groups. Two dose and three dose levels will be evaluated. Adult (aged 18-49 years), adolescents (aged 6-17 years), infant subjects (aged 7-71 months) and infant subjects (aged 2-6 months) will receive intramuscular (IM) injection on Days 0 and 28. Infant subjects (aged 2-6 months) subjects will receive intramuscular (IM) injection on Days 0 , 28 and 56. Three dose subgroups (low dose, medium dose and high dose were included in each age group. To maintain blindness in the trial, subjects were randomized in a 3:1 ratio to receive different dosages of the vaccine group or placebo group. In the analysis, the placebo subjects of the same age group were combined to ensure that the analysis ratio of the experimental vaccine group to the placebo group is 1:1. Therefore, 24 subjects in the experimental vaccine group and 8 subjects in the placebo group were chose in each dose group. Subjects were randomized to receive different dosages of the vaccine or placebo. Vaccination was performed in the adult group first, then on the adolescents, and on the infants last. Within each age group, dose-escalation with the principle from low to high dosage.

ELIGIBILITY:
Inclusion Criteria:

1. 2 months old to 49 years old, healthy resident, excluding the following:

   * Congenital malformations, developmental disorders, genetic defects, severe malnutrition and other conditions；
   * Have Congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus Erythematosus (SLE) , juvenile Rheumatoid Arthritis, or other autoimmune diseases；
   * History of Cerebral Palsy, seizures, mental illness.
2. I and/or my guardian voluntarily participate and sign an informed consent form, and can follow the requirements of the clinical trial protocol;
3. Have never received oral rotavirus live attenuated vaccine.

Exclusion Criteria:

* First dose exclusion criteria:

  1. Armpit temperature >37.0℃ before vaccination；
  2. Subjects with history of intussusception or suffering from intussusception；
  3. Subjects with history of convulsions and convulsions; history of epilepsy, mental illness and their family history；
  4. Subjects with history of allergy to vaccination；
  5. Acute attacks of various acute diseases (fever) or chronic diseases within 3 days before receiving the study vaccine；
  6. Subjects receiving immune enhancement or immunosuppressive therapy within 3 months (continuous oral or infusion for more than 14 days)；
  7. Subjects vaccinated with live attenuated vaccine within 14 days and other vaccines within 7 days before vaccination；
  8. Subjects with history of coagulation dysfunction (e.g. Coagulation factor deficiency, coagulation disease);
  9. Subjects with primary and secondary immunocompromised (history of thyroid, pancreas, liver, spleen resection, or need for treatment for thyroid disease in the past 12 months)；
  10. Subjects with abnormal blood biochemistry, blood routine, and urine routine related indicators that have clinical significance* before vaccination；
  11. Subjects who are currently or plan to participate in other clinical studies;
  12. According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

      Note*: The criterion of no clinical significance is "the laboratory test value between the upper limit (ULN) or lower limit (LLN) of the reference value range and the grade 1 adverse event" as judged by the doctor to have no clinical significance.
* In addition to the general exclusion criteria, specific subjects should also follow the following exclusion criteria.

（1）18-49-year-old women who have plans to become pregnant within the past 2 months or are pregnant or are breastfeeding； （2）Positive pregnancy test of female subjects of childbearing age； （3）18-49-year-old adults with hypertension that cannot be controlled by drugs (on site measurement: systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg)； （4）24-month-old infant subjects with a history of dystocia, suffocation rescue, neurological damage； （5）24-month-old baby subjects are born prematurely (delivered after the 37th week of pregnancy), low weight (birth weight for girls <2300g, boys <2500g).

-Exclusion criteria for follow-up needle:

1. Subjects with serious adverse reaction after the previous vaccination;
2. For the subjects who are newly discovered or newly appeared after the first vaccination that do not meet the selection criteria or meet the first exclusion criteria, the investigator will determine whether the subjects continue to participate the clinical trial;
3. Subjects vaccinated with other rotavirus vaccines other than the research vaccine during the study period;
4. Other exclusion reasons considered by the researcher.

Ages: 2 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Safety index-incidence of adverse reactions/events | 0-30 minutes after the first dose vaccination
  Incidence of adverse reactions/events after the first dose vaccination.
Safety index-incidence of adverse reactions/events | 0-30 minutes after the second dose vaccination
  Incidence of adverse reactions/events after the second dose vaccination.
Safety index-incidence of adverse reactions/events | 0-30 minutes after the third dose vaccination
  Incidence of adverse reactions/events after the third dose vaccination.
Safety index-incidence of abnormal blood biochemistry assessment | Day 4 after the first dose vaccination
  Incidence of abnormal blood biochemistry assessment at Day 4 after the first dose vaccination, except children aged Month 2-71
Safety index-incidence of abnormal blood routine assessment | Day 4 after the first dose vaccination
  Incidence of abnormal blood routine assessment at Day 4 after the first dose vaccination, except children aged Month 2-71
Safety index-incidence of abnormal urine routine assessment | Day 4 after the first dose vaccination
  Incidence of abnormal urine routine assessment at Day 4 after the first dose vaccination, except children aged Month 2-71
Safety index-incidence of abnormal blood biochemistry assessment | Day 4 after the second dose vaccination
  Incidence of abnormal blood biochemistry assessment at Day 4 after the second dose vaccination, except children aged Month 2-71
Safety index-incidence of abnormal blood routine assessment | Day 4 after the second dose vaccination
  Incidence of abnormal blood routine assessment at Day 4 after the second dose vaccination, except children aged Month 2-71
Safety index-incidence of abnormal urine routine assessment | Day 4 after the second dose vaccination
  Incidence of abnormal urine routine assessment at Day 4 after the second dose vaccination, except children aged Month 2-71
Safety index-incidence of abnormal blood biochemistry assessment | Day 4 after the third dose vaccination
  Incidence of abnormal blood biochemistry assessment at Day 4 after the third dose vaccination, except children aged Month 2-71
Safety index-incidence of abnormal blood routine assessment | Day 4 after the third dose vaccination
  Incidence of abnormal blood routine assessment at Day 4 after the third dose vaccination, except children aged Month 2-71
Safety index-incidence of abnormal urine routine assessment | Day 4 after the third dose vaccination
  Incidence of abnormal urine routine assessment at Day 4 after the third dose vaccination, except children aged Month 2-71
Safety index-incidence of adverse reactions/events | Day 0 to7 after the first dose vaccination
  Incidence of adverse reactions/events after the first dose vaccination.
Safety index-incidence of adverse reactions/events | Day 8 to30 after the first dose vaccination
  Incidence of adverse reactions/events after the first dose vaccination.
Safety index-incidence of adverse reactions/events | Day 0 to7 after the second dose vaccination
  Incidence of adverse reactions/events after the second dose vaccination.
Safety index-incidence of adverse reactions/events | Day 8 to30 after the second dose vaccination
  Incidence of adverse reactions/events after the second dose vaccination.
Safety index-incidence of adverse reactions/events | Day 0 to7 after the third dose vaccination
  Incidence of adverse reactions/events after the third dose vaccination.
Safety index-incidence of adverse reactions/events | Day 8 to30 after the third dose vaccination
  Incidence of adverse reactions/events after the third dose vaccination.
Safety index-incidence of serious adverse events | From the beginning of the vaccination to 6 months after the last vaccination completed
  Occurrence of serious adverse reactions/events after vaccination.

SECONDARY OUTCOMES:
Immunogenicity index-seroconversion rates of neutralizing antibody | Day 28 after the second dose vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rates of neutralizing antibody | Day 28 after the third dose vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4-fold increase from baseline.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | Day 28, 90, 180 after the second dose vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | Day 28, 90, 180 after the third dose vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.

OTHER OUTCOMES:
Immunogenicity index-seroconversion rates of IgA antibody | Day 28 after the second vaccination
  IgA antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rates of IgA antibody | Day 28 after the third dose vaccination
  IgA antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4-fold increase from baseline.
Immunogenicity index-geometric mean titer (GMT) of IgA antibody | Day 28, 90, 180 after the second dose vaccination
  IgA antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean titer (GMT) of IgA antibody | Day 28, 90, 180 after the third dose vaccination
  IgA antibody assay will be performed using the ELISA method.
Immunogenicity index-seroconversion rates of IgG antibody | Day 28 after the second dose vaccination
  IgG antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rates of IgG antibody | Day 28 after the third dose vaccination
  IgG antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4-fold increase from baseline.
Immunogenicity index-geometric mean titer (GMT) of IgG antibody | Day 28, 90, 180 after the second dose vaccination
  IgG antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean titer (GMT) of IgG antibody | Day 28, 90, 180 after the third dose vaccination
  IgG antibody assay will be performed using the ELISA method.
Cellular immune responses of lymphocytes | Day 14 after the second vaccination
  Lymphocytes (NK cells, B lymphocytes and T lymphocyte) responses of children aged 7-71 months will be measured using Flow cytometry.
Cellular immune responses of cytokines | Day 14 after the second vaccination
  Cytokines (IL-2, IL-4, IL-6, IL-10, TNF - α and IFN - γ) responses of children aged 7-71 months will be measured using ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun Li, Ph.D, Study Chair — Chinese Academy of Medical Sciences
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Zhenzhou, Henan, China

REFERENCES:
- [Derived] Wu JY, Zhang W, Pu J, Liu Y, Huang LL, Zhou Y, Gao JM, Tan JB, Liu XL, Yang J, Lin XC, Feng GW, Yin N, Chen R, Hu XQ, Yi S, Ye J, Kuang XJ, Wang Y, Zhang GM, Sun MS, Wang YX, Hu ZY, Yang JS, Li HJ. A randomized, double-blind, placebo-controlled phase I clinical trial of rotavirus inactivated vaccine (Vero cell) in a healthy adult population aged 18-49 years to assess safety and preliminary observation of immunogenicity. Vaccine. 2024 Jul 25;42(19):4030-4039. doi: 10.1016/j.vaccine.2024.05.014. Epub 2024 May 24. PMID 38796326